CLINICAL TRIAL: NCT00272857
Title: Gene Transfer From Patients With Fanconi Anemia, Genotype A: A Pilot Study
Brief Title: Bone Marrow Cell Gene Transfer in Individuals With Fanconi Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, David Williams, Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 382; R01HL081499 (NIH); CCHMCEH002 (Other Grant/Funding Number: CCHMC); R01HL081499-01A1 (NIH)
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental)
  Interventions: Genetic: Retrovirus Construct

INTERVENTIONS:
Genetic: Retrovirus Construct — This study will use an experimental gene transfer procedure performed in a laboratory to insert a new FA gene into the participant's bone marrow cells. The gene-corrected bone marrow cells will then be re-infused into the participant and participants will be observed for successful gene transfer

SUMMARY:
Fanconi anemia (FA) is a disease that affects an individual's bone marrow. It is caused by a defective gene in the bone marrow cells that produce various types of blood cells. Individuals with FA may experience fatigue, bleeding, and increased infections. The purpose of this study is to evaluate the safety and effectiveness of a gene transfer procedure in generating new, healthy cells in individuals with FA.

DETAILED DESCRIPTION:
FA is a rare, inherited disease that is caused by a gene defect and that primarily affects an individual's bone marrow, resulting in decreased production of blood cells. The lack of white blood cells affects an individual's ability to fight infections, the lack of platelets may result in bleeding, and the lack of red blood cells usually leads to anemia. FA is typically diagnosed in childhood, and there is a high fatality rate. Bone marrow transplants are one common treatment for FA. However, there are many risks associated with transplantation, including rejection of the transplanted cells and graft-versus-host disease, a serious side effect in which donor cells attack the recipient's tissues. This study will use an experimental gene transfer procedure performed in a laboratory to insert a new FA gene into the participant's bone marrow cells. The gene-corrected bone marrow cells will then be re-infused into the participant and participants will be observed for successful gene transfer. The purpose of this study is to evaluate the safety and effectiveness of the FA gene transfer procedure and to determine the ability of the gene-corrected cells at generating new, healthy blood cells in individuals with FA.

This study will enroll individuals with FA. Participants will be required to have the initial bone marrow transfer procedure performed at Cincinnati Children's Hospital, but will be allowed to see their own doctor for the majority of study visits. Participants will first attend a screening visit, which will include a physical exam, blood draw for laboratory testing, and a bone marrow biopsy. Bone marrow cells will be collected from eligible participants and sent to a laboratory for the FA gene transfer procedure. Several days later, the gene-corrected cells will be re-infused back into the participants via an intravenous catheter. Side effects will be closely monitored for 12 hours following the procedure and participants may be required to spend an overnight in the hospital. Following discharge from the hospital, participants will be required to stay in the Cincinnati area for 3 days to undergo daily evaluations and physical examinations. Participants will continue to be followed very closely for the first year after cell re-infusion. Study visits will be held weekly for the first 3 weeks, and then every 3 months for the remainder of the year. Visits will include physical examinations, blood collection, and liver function testing. Bone marrow testing will occur at Months 3, 6, and 12. Follow-up visits will occur yearly for up to 15 years and will include blood collection, a physical exam, and review of medical history.

ELIGIBILITY:
Inclusion Criteria:

* FA, as determined by a positive test for increased sensitivity to chromosomal breakage with mitomycin C or diepoxybutane
* FA complementation group A, as determined by somatic cell hybrids or molecular characterization; transduction of peripheral blood or bone marrow cells with the complementation group of specific retrovirus used in this study must demonstrate correction of mitomycin C sensitivity or cell cycle arrest
* Weighs at least 7.5 kg
* Normal cytogenetics on bone marrow within 3 months of study entry
* A minimum of 2 x 10(6) CD34+ cells/kg after CD34+ selection of the harvested bone marrow or mobilized peripheral blood product must be available to proceed with thaw (if cryopreserved) and transduction
* Human leukocyte antigen (HLA) typing with initial donor limited search results that indicate a potentially acceptable matched unrelated donor in the National Marrow Donor Program database

Exclusion Criteria:

* Cancer
* Clonal cytogenetic abnormality on bone marrow or peripheral blood karyotype within 3 months of study entry
* Myelodysplastic syndrome based on the FAB classification including:

  1. Refractory anemia with ringed sideroblasts (RARS)
  2. Refractory anemia with excess blasts (RAEB)
  3. RAEB in transformation (RAEB-T)
  4. Chronic myelomonocytic leukemia (CMML) (myelodysplastic changes in greater than two cell lines, refractory anemia alone, or aplastic anemia with dysplastic changes are permitted)
* Positive baseline screening result for both of the following:

  1. Detection of Fanconi A proviral sequences by polymerase chain reaction (PCR) analysis
  2. Detection of replication competent retrovirus by repeat testing by PCR of gibbon ape leukemia virus (GALV) envelope sequence or a positive S+L- assay
* Pregnant or breastfeeding; women of childbearing potential who are enrolled will be advised that the drug may cause birth defects and will be required to use an acceptable form of contraception
* Concurrent enrollment in any other study using an investigational agent, excluding androgens and thyroxine
* Physical or emotional status that would prevent informed consent, protocol compliance, or adequate follow-up with participant or legal guardian
* Participants for whom an acceptable HLA identical matched sibling donor (HLA A, B, DRB1; 6/6 match) has been identified (HLA typing of normal siblings must be documented)

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2004-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Safety of gene transfer methods | 3months, 6 months and yearly up to 15 years post gene transfer
Short-term and long-term engraftment of gene-corrected autologous hematopoietic cells (all measured at Year 1) | 3months, 6 months and yearly up to 15 years post gene transfer

SECONDARY OUTCOMES:
Frequency and function of the integrated recombinant Fanconi vector | 3months, 6 months and yearly up to 15 years post gene transfer
Efficiency of engraftment of multilineage gene corrected clones | 3months, 6 months and yearly up to 15 years post gene transfer
Lineage contribution and longevity of molecularly distinguishable gene marked clones | 3months, 6 months and yearly up to 15 years post gene transfer
Development of myelodysplastic syndrome or overt leukemia (all measured at Year 1) | 3months, 6 months and yearly up to 15 years post gene transfer

CONTACTS AND LOCATIONS:
Overall Officials: Franklin O. Smith, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly PF, Radtke S, von Kalle C, Balcik B, Bohn K, Mueller R, Schuesler T, Haren M, Reeves L, Cancelas JA, Leemhuis T, Harris R, Auerbach AD, Smith FO, Davies SM, Williams DA. Stem cell collection and gene transfer in Fanconi anemia. Mol Ther. 2007 Jan;15(1):211-9. doi: 10.1038/sj.mt.6300033. PMID 17164793